CLINICAL TRIAL: NCT06193356
Title: Detection of Endoscopic Resection Scars and Delineation of Recurrence Amongst Non-experts is Less Accurate Than Experts But Trainable in a Short Learning Intervention
Brief Title: Detection of Endoscopic Resection Scars and Delineation of Recurrence is Trainable
Acronym: SCAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2024-0133 - ID16649
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Polyp; Colorectal Cancer
Keywords: endoscopy; advanced imaging; post-colonoscopy colorectal cancer; Colorectal polypectomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A survey containing 15 High Definition - White Light (HD-WL) and Narrow Band Imaging (NBI) images, a learning intervention on detection of RRA (LT), then another set of 15 images was circulated to a mailing list of the GIEQs (Gastrointestinal Endoscopy Quality and Safety) foundation. Each image contained the same questions: Is this a resection scar? Is there RRA? What is your level of confidence? Information on the participant was obtained: number of EMRs performed, grade (consultant vs trainee) and years of experience. Comparisons were made to expert opinion derived at a consensus meeting of the senior authors regarding the appearances of the scars using the approach set out in Desomer et al. 2017.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre learning tool (No Intervention): Assessment of endoscopic images prior to a learning tool about scars and recurrence
- post learning tool (Experimental): Assessment of endoscopic images after a learning tool about scars and recurrence
  Interventions: Other: Learning tool

INTERVENTIONS:
Other: Learning tool — Video based learning tool about detection of endoscopic resection scars and recurrence.
  Arms: post learning tool

SUMMARY:
Colorectal cancer is prevented by colonoscopy and polypectomy. Failure to recognize the endoscopic resection scar after Endoscopic Mucosal Resection (EMR) risks unrecognized recurrent or residual adenoma (RRA), which may propagate into post-colonoscopy colorectal cancer. Expert series suggest scar recognition and interrogation is well performed with a high negative predictive value of endoscopic imaging vs histopathology. In this study the authors will investigate the performance of endoscopic imaging in detecting RRA at an endoscopic resection scar amongst general endoscopist and the impact of a learning intervention on recognition of RRA.

After consent is given, the participant will open the online survey and fill this in.

First the participant will be asked to create a pseudonym (name+year of birth) and fill in their demographical information (Grade, years in current role, colonoscopy experience, experience of colonic tissue resection, country of employment

The first 15 pictures will be shown prior to a learning intervention. For each picture the same questions will be asked:

* Is this an endoscopic resection scar?
* Based on this image does the scar demonstrate evidence of residual or recurrent adenoma (RRA)?
* What is your level of confidence?
* If the scar shows RRA, how would you treat it? (skip if you feel no RRA).
* If the scar does not show RRA do you feel there is another diagnosis? After the first 15 pictures a video-based learning tool will be shown on detection of RRA.

After the learning tool 15 different pictures will be shown, the same questions will be asked. All responses will be collected by the investigators. Statistical analysis will be performed using visual studio code (Microsoft, Redmond, USA) Images will be selected from the 'Australian Colonic LSL Endoscopic Resection Study' (ACE) database, which is an international multicentre registry of images and videos for retrospective analysis of colonic lesions. Images, videos, procedural information, and histopathological data are stored on a secure online web portal after written informed consent of every participating patient.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists of any experience level

Exclusion Criteria:

* non consenting adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Performance of detecting a recurrence at an endoscopic resection scar. | 2 years
  Performance of detecting a recurrence at an endoscopic resection scar.

SECONDARY OUTCOMES:
Performance of a learning tool in improving detection of recurrence at an endoscopic resection scar | 2 year
  Performance of a learning tool in improving detection of recurrence at an endoscopic resection scar
Difference in performance of detecting a recurrence at an endoscopic resection scar between endoscopists with different experience level | 2 year
  Difference in performance of detecting a recurrence at an endoscopic resection scar between endoscopists with different experience level
Performance of a learning tool in improving detection of recurrence at an endoscopic resection scar compared between endoscopists with different experience level | 2 year
  Performance of a learning tool in improving detection of recurrence at an endoscopic resection scar compared between endoscopists with different experience level

CONTACTS AND LOCATIONS:
Overall Officials: David J Tate, PhD, Principal Investigator — UZ Ghent
Locations (1):
- UZ Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers